CLINICAL TRIAL: NCT00058604
Title: Autologous EBV Specific CTLs for Prophylaxis and Therapy of EBV Lymphoma Post Solid Organ Transplant
Brief Title: Prevention and Treatment of Epstein-Barr Virus (EBV) Lymphoma Following a Solid Organ Transplant Using EBV Specific Cytotoxic T Lymphocytes (CTLs).
Acronym: EUCLID
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor/Director Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H9454; Euclid; NCT00607698 (obsolete NCT alias)
Record Dates: First submitted 2003-04-08; First posted 2003-04-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Epstein-Barr Virus Infections; Lymphoproliferative Disorders
MeSH Terms: conditions — Epstein-Barr Virus Infections; Lymphoproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Each patient will receive a Biological/Vaccine Intravenous injection of EBV specific CTLs
  Interventions: Biological: Intravenous injection of EBV specific CTLs

INTERVENTIONS:
Biological: Intravenous injection of EBV specific CTLs — Each patient will receive injections of 2x10e7 , 5x10e7 , or 10e8 CTLs/m2 via IV injection. 6 weeks = 1 course

SUMMARY:
Patients who may have been infected with EBV (Epstein-Barr Virus) before or after the time of their transplant have a higher risk of developing Lymphoproliferative Disease (LPD) or may already have a form of this disease.

This research study uses Epstein Barr virus (EBV) specific cytotoxic T lymphocytes (CTLs). These cells have been trained to attack and kill (cytotoxic) EB virus infected cells.

We make these cells from the patients blood by first growing an EBV infected B cell line by infecting the blood with an EBV virus called B-95. We then treat these EBV infected B cells with radiation so they cannot grow and use them to stimulate T cells. This stimulation will train the T cells to kill EBV infected cells. We will then test the T cells to make sure they kill the EBV infected cells.

The purpose of this study is to find the largest safe dose of EBV specific CTLs, to learn what the side effects are, and to see whether this therapy might help prevent or cure EBV related cancers in solid organ transplant patients

DETAILED DESCRIPTION:
Participation in this study will be for one year. Patients will receive this treatment either while in hospital or in the outpatient clinic. Each patient will be entered into one of three different dosing schedules being evaluated. Three to six patients will be evaluated on each dosing schedule. Escalation will continue until unacceptable side effects are seen.

First, patients will be given Tylenol (for any aches/pains) and Benadryl (for any minor allergic reactions such as itching/rash). This is called premedication. Next, the T cells will be injected into the patients' vein (intravenously) over approximately 10 minutes. Patients will be closely watched during this time to make sure they do not experience any bad effects such as an allergic reaction. If the patient does not respond to the T cells or if during follow-up examinations evidence of relapse is shown, the patient may receive another (higher) dose of T cells approximately six weeks after their first injection. Patients may decide NOT to continue to receive this therapy (receive further injections), however, the follow-up period will still be for one year.

Each patient will be seen every two weeks in the clinic or contacted every two weeks by the research nurse or other member of the research team, for six weeks after the injection(s). They will then be seen or contacted monthly for 3 months and then once every three months for one year and again if relapse occurs or is suspected.

To learn more about the way the T cells are working and how long they last in the body, 40 mls (8 teaspoonfuls) of blood will be taken once before the injection of T-cells, every two weeks for 6 weeks after the injection, monthly for 3 months and then every 3 months for 1 year. This amount of blood will be less for small patients. We will also take another blood sample from the patient if relapse is suspected. Each patient will need to have a physical examination by their physician to check on their progress.

Additionally, before the injection of T-cells, once every two weeks after the injection for 6 weeks and once every month for 3 months and then once every 3 months for one year and again if relapse occurs or is suspected we will obtain a blood sample from the patient to evaluate for transplant rejection. The amount of blood that we will take will be 3-5 mls (1/2 to 1 teaspoon). If the patient has received a heart transplant they will also be asked to have other tests such as an ultrasound or tomography (similar to an x-ray) done to help with this evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients falling into one of the following categories:

  * Organ transplant recipients at high risk of developing LPD:
  * EBV seronegative recipients
  * Organ transplant recipients receiving OKT3 for immunosuppression
* Organ transplant recipients with evidence of LPD
* Organ transplant recipients with EBV DNA level >1,000 copies
* Age <70 yrs old
* Signed informed consent obtained from patient/guardian
* CTLs available
* Performance status; ECOG £ 2
* Creatinine < 3X normal
* Bilirubin < 5X normal
* AST < 5X normal
* Has not received any other investigational cellular therapies within the past 30 days.

Exclusion criteria:

* Patients with a severe intercurrent infection
* Patients with life expectancy of less than 6 weeks
* Patients receiving supplemental oxygen.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Generate autologous, EBV-specific, cytotoxic T cell lines (CTLs) from individuals receiving or having received a solid organ transplant (SOT). | pre-treatment
Administer autologous, EBV-specific CTLs to patients, to determine the safety of intravenous injections in these individuals | 1 year
Evaluate the antiviral and immunological efficacy of the infused CTLs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas